CLINICAL TRIAL: NCT01400750
Title: Prospective Randomized Trial Comparing Oral Ciproxin Plus Inhaled Colistin With Tobramycin for Inhalation for Eradication of P Aeruginosa Infection in Children With Cystic Fibrosis.
Brief Title: Comparison of 2 Treatment Regimens for Eradication of P Aeruginosa Infection in Children With Cystic Fibrosis
Acronym: CCTOBI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Prof M Proesmans, University Hospital Leuven, dep of pediatrics
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MP1
Record Dates: First submitted 2011-07-18; First posted 2011-07-22 (Estimated); Last update posted 2011-08-04 (Estimated); Status verified 2011-07

CONDITIONS: Cystic Fibrosis
Keywords: cystic fibrosis- P aeruginosa- eradication-child
MeSH Terms: conditions — Cystic Fibrosis | interventions — Ciprofloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ciproxin-inhaled Colistin (Active Comparator): oral ciprofloxacin (30mg/kg/day) plus inhaled colistimethate sodium (Colistineb® 2x2 mill U daily) for 3 months
  Interventions: Drug: oral ciprofloxacin plus inhaled colistin
- Tobramycine for inhalation (TIS) (Active Comparator): tobramycin inhalation solution (TOBI® 2x300 mg) for 28 days
  Interventions: Drug: TOBI

INTERVENTIONS:
Drug: oral ciprofloxacin plus inhaled colistin — oral ciprofloxacin (30mg/kg/day divided in 2 doses) for 3 months (CC) plus inhaled colistimethate sodium(Colistineb® 2x2 mill U daily)
  Other Names: Ciproxin ® - ciprofloxacin; Colistineb ®
  Arms: Ciproxin-inhaled Colistin
Drug: TOBI — tobramycin inhalation solution (TOBI® 2x300 mg) for 28 days
  Other Names: TOBI® - tobramycin inhalation solution (TIS)
  Arms: Tobramycine for inhalation (TIS)

SUMMARY:
Treatment of new Pseudomonas aeruginosa (Pa) infection in cystic fibrosis (CF) can postpone chronic infection. Aim of the study: compare 2 Pa eradication regimens in children with new Pa infection.

DETAILED DESCRIPTION:
Methods: CF children (0-18 years) with a new isolation of Pa from the airway were randomized to tobramycin inhalation solution (TOBI® 2x300 mg for 28 days) (TIS) or inhaled colistimethate sodium (Colistineb® 2x2 mill U daily) plus oral ciprofloxacin (30mg/kg/day) for 3 months (CC). The primary outcome was eradication at end of treatment. Secondary outcome parameters were time to Pa relapse, total and Pa specific IgG, FEV1, BMI and Pa status.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of CF (clinical signs consistent with CF and a sweat chloride > 60 mEq/l by quantitative pilocarpine iontophoresis and/or two CF causing mutations identified)
* age 0 to 18 years old at time of inclusion
* 'First' or 'new Pa infection' defined as 'first Pa isolation ever' or 'isolation of Pa from the airway (sputum, throat swab or BAL) after a Pa free interval of at least 6 months and documented with at least 3 negative cultures'.

Exclusion Criteria:

* chronic Pa infection defined according to the Leeds criteria[17]
* pulmonary exacerbation needing IV AB treatment at time of new Pa isolate
* Pa isolation at time of CF diagnosis
* patient already on an antipseudomonal antibiotic
* interval between positive culture and start of treatment > 4 weeks.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 61 (Actual)
Dates: Start 2001-08; Primary Completion 2010-08 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Pseudomonas aeruginosa eradication at the end of the treatment. | end of study drug treatment ie 3 months for CC and at 1 months for TIS
  sucessful eradication is defined as negative airway culture for P aeruginosa and end of study drug which is after 3 months for ciproxin-colistin (CC) and after 1 months for tobramycin for inhalation (TIS)

SECONDARY OUTCOMES:
P aeruginosa eradication at 6 months after study entry | 6 months
  negative airway cultures for P aeruginosa up to 6 months after start of study drug
time to new Pa positive culture (= relapse) | 1 year
  Time to first new P aeruginosa positive airway culture (expressed in months starting from end of study drug)
change from baseline FEV1% pred, IgG z score, BMI z score was followed | 1 year
  Evolution of lung function (expressed as FEV1% pred), total IgG and nutritional status (expressed as BMI z score) from start of study up to 1 year
Antibody titer for specific anti Pseudomonas antibodies | 1 year
  Pa antibodies (ELISA St Ag 1-17 )were measured at baseline and at 1 year follow-up
P aeruginosa infection status | 1 year
  P aeruginosa infection status was reported as 'Free off', 'Intermittent' or 'Chronic' according to the Leeds criteria after 1 and 2 years.
  (ref Leeds criteria: Lee TW, Brownlee KG, Conway SP, et al. Evaluation of a new definition for chronic Pseudomonas aeruginosa infection in cystic fibrosis patients. J Cyst Fibros 2003;2(1):29-34)
P aeruginosa infection status | 2 years
  P aeruginosa infection status was reported as 'Free off', 'Intermittent' or 'Chronic' according to the Leeds criteria after 1 and 2 years.
  (ref Leeds criteria: Lee TW, Brownlee KG, Conway SP, et al. Evaluation of a new definition for chronic Pseudomonas aeruginosa infection in cystic fibrosis patients. J Cyst Fibros 2003;2(1):29-34)

CONTACTS AND LOCATIONS:
Overall Officials: Marijke J Proesmans, MD, PhD, Principal Investigator — Dep pediatrics University Hospital Leuven Belgium
Locations (1):
- Department of pediatrics, CF center Uuiversity Hospital Leuven, Leuven, Belgium

REFERENCES:
- [Result] Langton Hewer SC, Smyth AR. Antibiotic strategies for eradicating Pseudomonas aeruginosa in people with cystic fibrosis. Cochrane Database Syst Rev. 2009 Oct 7;(4):CD004197. doi: 10.1002/14651858.CD004197.pub3. PMID 19821321